CLINICAL TRIAL: NCT03114553
Title: Integration of Family Health History Data Into a Singaporean Healthy Population Cohort Database to Understand the Associations Between Family Health History and Genomics
Brief Title: Family History in a Singaporean Healthy Population
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00079760
Record Dates: First submitted 2017-04-11; First posted 2017-04-14 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: All
Keywords: family health history; prevention; genetic risk; clinical decision support
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: MeTree — Software program collecting family health history and generating clinical decision support for risk-based preventive care
  Other Names: patients in the database have already had biologic specimens for genetic analysis

SUMMARY:
The purpose of this study is to better understand the linkages between family health history (FHH) and genomics in a Singaporean population. Secondly this study will evaluate the facilitators and barriers to implementation of a family history collection and risk assessment tool within a Singaporean population.

DETAILED DESCRIPTION:
This study is a collaboration between Duke University School of Medicine Center for Applied Genomics and Precision Medicine (CAGPM) and the National Heart Center of Singapore (NHCS) and SingHealth Duke-NUS Center for Precision Medicine (PRISM). The NHCS study, Molecular and Imaging Studies of Cardiovascular Health and Disease ("Biobank study") is collecting genomic, clinical, and environmental data on a large cohort of healthy Singaporean volunteers. Data from the Biobank study is being deposited into a large healthy population cohort database, SPECTRA, organized under PRISM. The investigators will collaborate with the NHCS Biobank study and PRISM to integrate the Duke family history risk assessment platform, MeTree, into the data collection of the Biobank study cohort for in-depth analyses of FHH and genomic associations as well as exploration of the feasibility of MeTree implementation into the Singaporean clinical context. The Biobank study is a prospective observational study. It has already enrolled 1,000 subjects and will continue enrollment over the next year and possibly beyond. Previously enrolled subjects will be re-contacted for completion of MeTree as well as having future enrollees complete the tool prospectively. The investigators anticipate 5,000 subjects completing MeTree over a one-year period. The investigators will evaluate the feasibility and effectiveness of implementing MeTree in the larger Singaporean context. The investigators will assess implementation related outcomes- questions/problems people have when completing their family histories, how complete are the FHH entered, what types of risk are identified and what existing programs in Singapore are designed to manage that risk. The completion of this project will provide a significant amount of data to better understand the associations between FHH and genomic data within a healthy Asian population. It also will result in a better understanding of an appropriate implementation strategy for MeTree within the Singaporean clinical setting.

Specific Aim 1: To explore the correlation of genomic data and FHH within a healthy Asian population.

Specific Aim 2: To assess the clinical utility and appropriateness of a patient-entered FHH risk assessment tool within a Singaporean population.

Specific Aim 3: To create an implementation strategy for broader implementation of a patient-driven risk assessment tool in Singapore.

Duke University will be providing access to the MeTree Family Health History tool, storage of the PRISM participant data, participant and provider risk assessment reports, and education about the tool to PRISM study staff as needed. Duke University personnel will not be involved in any recruiting, consenting, or follow-up with study participants, but will have access to de-identified participant data housed in the MeTree research database in order to provide support for the study coordinators for participant account trouble-shooting and also to provide interim and final datasets to the PRISM statisticians. The MeTree research database currently sits on a DHTS server behind the Duke firewall, and is maintained and secure in accordance with Duke policy for patient data.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Singaporeans enrolled or eligible for enrollment in a local Biobank protocol

Exclusion Criteria:

-

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy Singaporean population
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2017-07-23 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Correlation of genomic data and family health history (FHH) within a healthy Asian population. | Baseline
  assess whether family history driven risk results correlate with findings on genetic results

SECONDARY OUTCOMES:
Clinical utility and appropriateness of a patient-entered FHH risk assessment tool within a Singaporean population | Baseline
  Determine whether US guideline driven risk assessment has any clinical value in Singapore
Facilitators and barriers to using systemic risk assessment tool in Singapore | Baseline
  Identify facilitators and barriers to using risk assessment tool in order to create a strategy for broader implementation of a patient-driven risk assessment tool in Singapore

CONTACTS AND LOCATIONS:
Overall Officials: Lori Orlando, MD, Principal Investigator — Associate Professor of Medicine
Locations (1):
- National Heart Centre of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu RR, Sultana R, Bylstra Y, Jamuar S, Davila S, Lim WK, Ginsburg GS, Orlando LA, Yeo KK, Cook SA, Tan P. Evaluation of family health history collection methods impact on data and risk assessment outcomes. Prev Med Rep. 2020 Mar 5;18:101072. doi: 10.1016/j.pmedr.2020.101072. eCollection 2020 Jun. PMID 32181122
- [Result] Bylstra Y, Lim WK, Kam S, Tham KW, Wu RR, Teo JX, Davila S, Kuan JL, Chan SH, Bertin N, Yang CX, Rozen S, Teh BT, Yeo KK, Cook SA, Jamuar SS, Ginsburg GS, Orlando LA, Tan P. Family history assessment significantly enhances delivery of precision medicine in the genomics era. Genome Med. 2021 Jan 7;13(1):3. doi: 10.1186/s13073-020-00819-1. PMID 33413596